CLINICAL TRIAL: NCT00002822
Title: RANDOMISED CLINICAL TRIAL OF IFOSFAMIDE, CARBOPLATIN AND ETOPOSIDE WITH MID-CYCLE VINCRISTINE (VICE) VERSUS STANDARD PRACTICE CHEMOTHERAPY IN PATIENTS WITH LIMITED STAGE SMALL CELL LUNG CANCER (SCLC) AND GOOD PERFORMANCE STATUS
Brief Title: Combination Chemotherapy Followed by Radiation Therapy in Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064998; MRC-LU21; EU-96019
Record Dates: First submitted 1999-11-01; First posted 2003-04-16 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2000-12

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer; extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Doxorubicin; Etoposide; Ifosfamide; Mesna; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: mesna
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug is a way to kill more tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effect of two combination chemotherapy regimens followed by radiation therapy in treating patients with small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival rate in patients with newly diagnosed small cell lung cancer and good performance status treated with an intensive regimen of ifosfamide/carboplatin/etoposide with mid-cycle vincristine (VICE) vs. standard chemotherapy followed, as feasible, by thoracic radiotherapy.
* Compare the adverse effects of treatment and quality of life (including psychological distress, physical status, and functional status and global quality of life) in these patients.
* Compare the Rotterdam Symptom Checklist vs. the EORTC QLQ-C30 and LC13 quality-of-life questionnaires in relation to compliance and ability to detect differences between treatments.

OUTLINE: This is a randomized study.

The first group receives standard combination chemotherapy with doxorubicin/cyclophosphamide/etoposide (ACE) or cisplatin/etoposide (PE) every 3 weeks for 6 courses.

The second group receives intensive combination chemotherapy with carboplatin/ifosfamide/etoposide on days 1-3 with vincristine on day 14 (VICE). Courses repeat every 4 weeks for 6 courses.

Patients in both groups are considered for thoracic radiotherapy beginning 4-5 weeks after the first day of the last course of chemotherapy.

Concurrent prophylactic antibiotics should be given. Patients who relapse may receive further treatment at the clinician's option.

Patients are followed monthly for 6 months, every 2 months for up to 1 year, every 3 months for up to 2 years, every 6 months for 5 years, and annually thereafter.

PROJECTED ACCRUAL: A total of 400 patients will be entered over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Microscopically proven small cell lung cancer

  * Diagnosis based on bronchial, mediastinal, pleural, lung, or lymph node biopsy, sputum cytology, or bronchial brushing or fine needle aspirate cytology
  * No pleural fluid cytology
* No prior therapy

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* WHO 0-2

Hematopoietic:

* WBC more than 3,000
* ANC more than 1,500
* Platelets more than 100,000

Hepatic/Renal:

* Alkaline phosphatase, aminotransferase, sodium, and LDH normal or no more than 1 of them abnormal
* Creatinine or urea normal
* Creatinine clearance or GFR more than 65 mL/min

Other:

* No clinical evidence of infection
* No prior or concurrent malignancy that interferes with protocol treatments or comparisons
* No other condition that contraindicates treatment
* Willing and able to complete quality-of-life questionnaires

  * Hospital Anxiety and Depression Scale, Rotterdam Symptom Checklist, and EORTC questionnaires completed prior to randomization

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 1996-03; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Girling, MD, Study Chair — Medical Research Council
Locations (1):
- Medical Research Council Clinical Trials Unit, London, England, United Kingdom

REFERENCES:
- [Result] Thatcher N, Qian W, Clark PI, Hopwood P, Sambrook RJ, Owens R, Stephens RJ, Girling DJ. Ifosfamide, carboplatin, and etoposide with midcycle vincristine versus standard chemotherapy in patients with small-cell lung cancer and good performance status: clinical and quality-of-life results of the British Medical Research Council multicenter randomized LU21 trial. J Clin Oncol. 2005 Nov 20;23(33):8371-9. doi: 10.1200/JCO.2004.00.9969. PMID 16293867
- [Result] Thatcher N, Qian W, Girling DJ: Ifosfamide, carboplatin and etoposide with mid-cycle vincristine (ICE-V) versus standard chemotherapy (C) in patients with small cell lung cancer (SCLC) and good performance status (PS): results of an MRC randomized trial (LU21). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2489, 619, 2003.